CLINICAL TRIAL: NCT06019260
Title: Open Versus Arthroscopic Assisted Treatment of Acute Acromioclavicular Joint Disruption Using Suture Button Device
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Adel Abdelmajeed, resident doctor, Assiut University
Other Study IDs: Acute AC Joint disruption
Record Dates: First submitted 2023-07-18; First posted 2023-08-31 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Acromioclavicular Joint Dislocation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group 1: open surgical repair using suture button device method in acute acromioclavicular joint disruption
- group 2: arthroscopic assisted treatment of acute acromioclavicular joint disruption using suture button device

SUMMARY:
Compare the clinical and radiological outcome between the arthroscopic and open surgical repair using suture button device method in cases with acute AC joint disruption

DETAILED DESCRIPTION:
Acromioclavicular (AC) joint dislocation is a common shoulder injury, especially among athletes and has an estimated incidence of 17% of all shoulder injuries and30%-50% of athletic shoulder injuries ,In most cases, these are caused by a direct fall on the ipsilateral shoulder tip. The indirect mechanism of injury with an extended arm is rare, The Rockwood classification system is currently used and based on the degree and direction of the disrupted anatomy of the AC joint.

Despite the high prevalence of this injury, there is no consensus about its optimal treatment. A variety of surgical procedures are described in the literature, such as an augmented suture with absorbable materials, stabilization with Kirschner (K)-wires in combination with or without additional wire loops, hook plates, or the Bosworth screw, but none can be considered the gold standard of operative AC joint stabilization, another treatment option was offered by the Tight Rope system, This technique was developed as a minimally invasive procedure in the management of AC dislocations. Because of its minimally invasive approach, it reduces soft tissue damage and yields better cosmetic results.9 Also, there is no need for reoperation to remove the hardware that might screws, or plates. Moreover, the complications of hardware failure, like breakage, dislocations, or bone fractures, are minimized

ELIGIBILITY:
Inclusion Criteria:

* Age of 16 to 60 years
* Definite radiographic diagnosis of isolated Rockwood type IIIb(unstable), IV and type v acromioclavicular joint dislocation
* Time from injury to operation < 3 weeks
* Patient with complete at least 12-month follow-up assessments

Exclusion Criteria:

* . Age outside the range

  * Open injury, old injury (≥ 3 weeks since injury)
  * Injury caused by other diseases (tendinitis, metabolic, et al.), concurrent shoulder osteoarthritis, arthropathy or any fracture
  * Any previous operation of the injured limb
  * Incomplete data or follow-up < 12 months

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients meeting the inclusion criteria and willing to take part in the study will be included investigators conducted an a priori test for sample size calculation using the G*Power 3.1.9.2 software. investigators assumed a CMS mean difference between the 2 groups of 16 points, a standard deviation of 20 points, an alpha of 0.05, and power (1 - b) of 80%; 21 subjects had to be included in each group. Our goal was to include 27 cases in each group to compensate for any lost subjects during the follow-up phase
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Radiological evaluation using the true anteroposterior view of the shoulder | preoperative, three month postoperative and six month postoperative
  Radiological evaluation using the true anteroposterior view of the shoulder and AC projection (10 cephalic tilt with the beam centered over the AC joint)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeong JY, Chun YM. Treatment of acute high-grade acromioclavicular joint dislocation. Clin Shoulder Elb. 2020 Sep 1;23(3):159-165. doi: 10.5397/cise.2020.00150. eCollection 2020 Sep. PMID 33330252
- [Background] Vijayan S, Kulkarni MS, Jain CP, Shetty S, Aroor MN, Rao SK. Bifocal Stabilisation of Acute Acromioclavicular Joint Dislocation using Suture Anchor and Temporary K-Wires: A Retrospective Analysis. Malays Orthop J. 2022 Nov;16(3):104-112. doi: 10.5704/MOJ.2211.016. PMID 36589364
- [Background] Bezruchenko S, Dolhopolov O, Yarova M, Luchko R, Mazevych V. Clinical Evaluation and Instrumental Diagnostics in Acute Acromioclavicular Joint Dislocation. Ortop Traumatol Rehabil. 2022 Feb 28;24(1):1-12. doi: 10.5604/01.3001.0015.7800. PMID 35297375
- [Background] Liu X, Huangfu X, Zhao J. Arthroscopic treatment of acute acromioclavicular joint dislocation by coracoclavicular ligament augmentation. Knee Surg Sports Traumatol Arthrosc. 2015 May;23(5):1460-1466. doi: 10.1007/s00167-013-2800-9. Epub 2013 Dec 10. PMID 24318508
- [Background] Lu D, Wang T, Hong JJ, Chen H, Sun LJ. Acute acromioclavicular joint dislocation treated with tightrope : Mini-open versus percutaneous stabilization. Acta Orthop Belg. 2019 Dec;85(4):406-411. PMID 32374229